CLINICAL TRIAL: NCT03528096
Title: Feasibility Study of Contactless 3D Video Assessment and 'Somnomat' Vestibular Stimulation Therapy in Childhood Rhythmic Movement Disorder
Brief Title: Vestibular Stimulation Therapy for Rhythmic Movement Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University of Southampton (Other); AIT Austrian Institute of Technology GmbH (Other); University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RMD-SOMNOMAT
Record Dates: First submitted 2018-05-04; First posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Sleep Related Rhythmic Movement Disorder (Disorder)
MeSH Terms: interventions — Sound

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant
Masking Description: Blinding of the participants is impossible, as the stimulation is easy to perceive and cannot be confused with a baseline night. Therefore, participants are informed about the character of the night (max. 5 minutes) before the moment of lights off. For safety reasons the experimenter that is present is also aware of the condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention night (Experimental): Vestibular stimulation, in the form of gentle rocking movements, is provided using the Somnomat B rocking bed. Stimulation is provided for the first 60 minutes of the night and for 10 minutes upon detection of symptoms. The stimulation frequency is in the range of 0.25-2 Hz.
  Interventions: Device: Somnomat B
- Baseline night (Sham Comparator): The sound of the moving bed is played back to the participant at the right sound intensity level.
  Interventions: Other: Sound

INTERVENTIONS:
Device: Somnomat B — Vestibular stimulation is provided using an innervated bed platform. This robotic device consists of a standard single bed, mounted on a moving mechanism. It was developed and produced by the ETH Zürich and approved for use in this study by Swissmedic.
  Arms: Intervention night
Other: Sound — Sound of the moving bed was recorded and played back during the baseline night.
  Arms: Baseline night

SUMMARY:
This study aims to a) investigate the feasibility of the detection of episodes of RMD using contactless 3D video analysis and customised analysis software and b) the use of vestibular stimulation as a therapy for childhood rhythmic movement disorder.

DETAILED DESCRIPTION:
Rhythmic movement disorder (RMD) is a childhood onset sleep disorder that is characterised by repetitive movements that involve large muscle groups, such as body rocking, rolling and head banging. These rhythmic movements are performed prior to and during sleep and as such can disturb sleep with clinical consequences. There is no standard measure to quantify the severity of rhythmic movements. 3D video offers a contactless method of achieving this without disrupting the child's sleep. Vestibular stimulation has a soothing effect and might be effective in promoting sleep. Furthermore, mild vestibular stimulation in the form of gentle rocking movements generated by the Somnomat device might function as a stimulation substitute for the child's RMD with therapeutic potential.

This study aims to a) investigate the feasibility of the detection of episodes of RMD using contactless 3D video analysis and customised analysis software and b) the use of vestibular stimulation as a therapy for childhood rhythmic movement disorder.

ELIGIBILITY:
Inclusion Criteria:

* RMD diagnosis based on ICSD III criteria or RMD suspected
* Typically developing
* Child and accompanying adult are legally allowed to enter Switzerland without a visa
* Both child and parent/legal guardian understand easy English or German

Exclusion Criteria:

* Moderate or severe learning disability
* Neurological disorder (incl. autism, epilepsy, medicinally treated ADHD)
* Currently using medication that influences sleep
* Known diseases of the vestibular system
* Self-reported sensitivity for motion sickness
* Body height > 1.95 m (due to the constraints of the setup)
* Body weight > 130 kg (due to the constraints of the setup)
* Flu, cold or other acute disease on study day that might influence measurements
* Pregnancy

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Effect of Therapy on Subjective Sleep Quality | 2 nights
  Difference in perceived sleep quality between baseline and intervention nights. Data is collected in the first hour after awakening using a questionnaire.
Reliability of Automatic Detection of Symptoms | 3 nights
  Episodes of rhythmic movement scored by an algorithm using 3D Video will be compared to the scoring of an expert

SECONDARY OUTCOMES:
Effect of Therapy on Objective Sleep Quality | 2 nights
  Sleep quality is determined based on 2D video recordings and compared between baseline and intervention nights.
Effect of Therapy on Symptoms | 2 nights
  Severity of symptoms is determined based on 2D video recordings. The number of episodes of rhytmic movement (count) and the duration of episodes (minutes) compared between baseline and intervention nights.
Preferred Stimulation Parameters | 1.5 hours
  Participants can try out different directions of movement (pitch or roll) and different movement frequencies between 0 and 2 Hz and choose their preferred settings (one direction + one frequency).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Riener, Prof. Dr., Principal Investigator — ETH Zürich
Locations (1):
- Sensory Motor Systems Lab, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gall M, Kohn B, Wiesmeyr C, van Sluijs RM, Wilhelm E, Rondei Q, Jager L, Achermann P, Landolt HP, Jenni OG, Riener R, Garn H, Hill CM. A Novel Approach to Assess Sleep-Related Rhythmic Movement Disorder in Children Using Automatic 3D Analysis. Front Psychiatry. 2019 Oct 16;10:709. doi: 10.3389/fpsyt.2019.00709. eCollection 2019. PMID 31681030